CLINICAL TRIAL: NCT04189146
Title: Inner Engineering Yoga Program on Short and Long Term Health Effects (ISHA-Impact): A Longitudinal Study
Acronym: ISHA-Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Director, Center for Anesthesia Research Excellence, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P000205
Record Dates: First submitted 2019-10-11; First posted 2019-12-06 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Mediation; Mood; Stress; Habits; Nicotine; Alcohol Consumption; Pain Intensity; Sleep; Mindfulness; Emotions; Anxiety; Depression
MeSH Terms: conditions — Negotiating; Habits; Alcohol Drinking; Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study only involves administration of electronic surveys at six different time points. These time points include: at the time of consent; after completing the Inner Engineering Online modules but before the in-person course begins; after the completion of the in-person (IECO) course; at 6 weeks; at 6 months and at 12 months. These surveys can take up to 15 minutes to complete. Electronic reminders will be sent to participants who have not completed these surveys within a week.
  Additionally, participants must complete a two-minute compliance survey at the end of each week for 6 weeks after IECO completion. After these 6 weeks, this same two-minute compliance survey will be sent monthly until the end of the year. This survey is an important component of our data analysis, because it collects information on the frequency and duration of their routine practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inner Engineering Intervention (Other): The intervention investigators propose for the study includes an Online Course with 7 modules, or a 10 hours long course, and a 1-2 day In-Person Course, in which participants will learn a simple 21 minute practice called Shambhavi Mahamudra Kriya, also known as Shambhavi Kriya.
  Interventions: Behavioral: Inner Engineering Intervention

INTERVENTIONS:
Behavioral: Inner Engineering Intervention — The intervention investigators propose for the study includes an Online Course with 7 modules, or a 10 hours long course, and a 1-2 day In-Person Course, in which participants will learn a simple 21 minute practice called Shambhavi Mahamudra Kriya, also known as Shambhavi Kriya.
  Shambhavi Kriya is a powerful and purifying energy technique incorporating the breath. This practice is said to align the participants system such that their body, mind and emotions function in harmony.

SUMMARY:
This study will include any participant who registered, and plans to attend the Inner Engineering In-Person Completion Course. In 2019, this course was offered in: Los Angeles in March, Philadelphia in April and Toronto & Dallas in November. This study has been involved in every IECO Course since 2019 and is still active today. Beginning in August 2021, investigators will recruit for the August Inner Engineering In-Person Completion Course. Investigators anticipate that this study can include up to 5,000 study participants. Participants would attend this course and complete the pre-modules regardless of whether or not they participate in this study.

DETAILED DESCRIPTION:
This study aims to enroll participants who have registered for the Inner Engineering in-person course. Briefly, this course is a 1-2 day in-person course, in which participants will learn a simple 21 minute practice called Shambhavi Mahamudra Kriya, also known as Shambhavi Kriya. Shambhavi Kriya is a powerful and purifying energy technique which incorporates the breath. This practice is said to align the body systems so that the body, mind and emotions function in harmony. More information about the course can be found on the ISHA foundation website: https://www.innerengineering.com/ieo-new/completion/.

Registrants for IECO are asked to complete a series of seven (7) online modules (IEO) prior to the start of the in-person course. The online series provides the participants with an opportunity to intellectually explore the basics of life using methods that are distilled from the essence of yogic sciences. The course imparts wisdom to manage the body, mind, emotions, and the fundamental life energy within.

Importantly, the course modules (IEO) and the in-person meeting (IECO) and subsequent meditation and yoga practices would occur regardless of whether or not a person decided to participate in the study. The only study procedure imparted includes requesting the participants to complete a series of surveys over a one-year period.

This study only involves administration of electronic surveys at six different time points. These time points include: at the time of consent; after completing the Inner Engineering Online modules but before the in-person course begins; after the completion of the in-person (IECO) course; at 6 weeks; at 6 months and at 12 months. These surveys can take up to 15 minutes to complete. Electronic reminders will be sent to participants who have not completed these surveys within a week.

Additionally, participants must complete a two-minute compliance survey at the end of each week for 6 weeks after IECO completion. After these 6 weeks, this same two-minute compliance survey will be sent monthly until the end of the year. This survey is an important component of our data analysis, because it collects information on the frequency and duration of their routine practice.

Participants can choose to either complete their baseline & post-IEO surveys only, or continue and complete Post IECO- 1 year follow up period. A break was incorporated because IEO & IECO are 2 separate events, and participants who chose to complete IEO may not necessarily complete IECO. This break ensures maximum participation.

This study will include participants who are registered and plan to attend any Inner Engineering Online & Inner Engineering Online Completion Course. This course is offered several times throughout the year and each course has several hundred participants. We anticipate we can collect data from up to 5,000 study participants and create a significant database of Inner Engineering practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have registered to take the Inner Engineer Online Course.
* Participants who have registered to take the Inner Engineer Completion Course.
* Participants must be able to read and understand English.

Exclusion Criteria:

* Participants who report living outside the United States at the time of enrollment.
* Participants < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Perceived Stress Levels | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The study aims to evaluate changes in perceived levels of stress in survey participants and the effect Inner Engineering has over them in long term. The investigators use a validated scale for this purpose named, Perceived Stress Scale (PSS). The scale measures the degree to which situations in participant's life are appraised as stressful. This is defined to be the key secondary outcome for the study. Higher scores are suggestive of more stress. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Mood Changes | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The study aims to evaluate changes in mood profiles affected by the Inner Engineering Online (IEO) over time. For evaluation of mood profiles the investigators use a validated scale named, Profile of Mood States (POMS). The scale measures different dimensions of mood swings over a period of time and calculates Total Mood Disturbances by performing a sub-scale analysis. The subscales defined include Tension, Depression, Anger, Fatigue, Confusion & Vigor. Higher scores are suggestive of poorer outcome. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.

OTHER OUTCOMES:
Habits of daily living | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose named, NHANES III. The scale measures the habits of daily living of an individual. This is a qualitative scale, and scoring is not done. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Nictoine Consumption | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use several validated scale for this purpose namely, NHANES III, Nicotine dependence, Negative Health Expectancies and Emotional Expectancies among others. The scales measure the nicotine dependence and aids in quantifying dependence which in turn aids in evaluating any change on the individual's perception after the Inner Engineering intervention. Higher scores suggest greater nicotine dependence. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Alcohol Consumption | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose namely, AUDIT. The scale measures the individual's dependence on alcohol and objectively quantifies dependence which in turn aids in evaluating any change on the individual's perception after the Inner Engineering intervention. A score of 8 or more is considered to be hazardous use of alcohol. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Pain Intensity | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose namely, Pain intensity & Pain interference scales. The scales measure the individuals' pain perception, and quantify the effects of the individuals' pain which in turn aids in evaluating any change on the individual's perception after the Inner Engineering intervention. higher scores suggestive of increased pain perception. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Sleep patterns & behavior | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose namely, Pittsburgh Sleep Quality Index (PSQI). The scale measure the individuals' sleep patterns & behavior and quantifies sleep quality which in turn aids in evaluating any change on the individual's sleep quality after the Inner Engineering intervention. Scores higher than 5 are suggestive of poor sleep quality. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Mindfulness | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose namely, Mindfulness Attention Awareness Scale (MAAS). The scale measures the individuals' ability for receptive awareness and attention to present. This aids in evaluating any change on the individual's awareness levels after the Inner Engineering intervention. Higher scores are suggestive of increased mindfulness and awareness. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Emotional health | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators use a validated scale for this purpose namely, PERMA profiler. The scale measures the 5 pillars of well-being (Positive emotions, engagement, relationship, meaning, accomplishment) along with negative emotions and health in the individual. Higher scores are suggestive of better outcomes. This aids in evaluating any change on the individual's awareness levels after the Inner Engineering intervention. Logistic regression analysis is performed on the outcome measures collected over the specified time-frame.
Anxiety | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators used the PROMIS (Anxiety-8) an 8-item validated instrument that assesses the severity of anxiety. Participants are asked on a scale of 1 (Never) to 5 (Always) on the frequency of occurrence of each negative experience. Overall score is computed based on sum from individual responses. A higher sum indicates greater anxiety.
Depression | The investigators collect these scores at the 6 pre-specified time points; i.e., at the time of consent; after completing the IEO modules but before conference; post conference completion; at 6 weeks; at 6 months and at 12 months.
  The investigators used the CES-D 20-item scale to assess depression. Each item is coded 1 "rarely or none of the time (less than 1 day)" to 4 "most or all of the time (5-7 days)." Scores range from 0 to 60, with high scores indicating greater depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyman SA, Shotwell MS, Michaels DR, Han X, Card EB, Morse JL, Weinger MB. A Survey Evaluating Burnout, Health Status, Depression, Reported Alcohol and Substance Use, and Social Support of Anesthesiologists. Anesth Analg. 2017 Dec;125(6):2009-2018. doi: 10.1213/ANE.0000000000002298. PMID 28991114
- [Background] Kato T. Development of the Sleep Quality Questionnaire in healthy adults. J Health Psychol. 2014 Aug;19(8):977-86. doi: 10.1177/1359105313482168. Epub 2013 May 29. PMID 23720542
- [Background] Shioata, M.N., D. Keltner, and O.P. John, Positive Emotion Dispositions Differntially Associatd with Big Five Personality and Attachement Style. The Journal of Positive Psychology, 2006. 1(2): p. 61-71.
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Ryan RM, Deci EL. On happiness and human potentials: a review of research on hedonic and eudaimonic well-being. Annu Rev Psychol. 2001;52:141-66. doi: 10.1146/annurev.psych.52.1.141. PMID 11148302
- [Background] Peterson CT, Bauer SM, Chopra D, Mills PJ, Maturi RK. Effects of Shambhavi Mahamudra Kriya, a Multicomponent Breath-Based Yogic Practice ( Pranayama), on Perceived Stress and General Well-Being. J Evid Based Complementary Altern Med. 2017 Oct;22(4):788-797. doi: 10.1177/2156587217730934. Epub 2017 Sep 22. PMID 29228793
- [Background] Muralikrishnan K, Balakrishnan B, Balasubramanian K, Visnegarawla F. Measurement of the effect of Isha Yoga on cardiac autonomic nervous system using short-term heart rate variability. J Ayurveda Integr Med. 2012 Apr;3(2):91-6. doi: 10.4103/0975-9476.96528. PMID 22707866
- [Background] Selvaraj, N., et al., Heart Rate Dynamics during Shambhavi Mahamudra - A Practice of Isha Yoga. Journal of Complementary and Inegrative Medicine, 2008. 5(1): p. 1-22.
- [Derived] Swaminathan A, DeSchryver B, Rayapuraju A, Barbaro J, Orui H, Subramaniam B, Reed PU. From strain to strength: a yearlong study on the transformative influence of inner engineering online program on mental well-being. Front Psychol. 2025 Feb 4;16:1436910. doi: 10.3389/fpsyg.2025.1436910. eCollection 2025. PMID 39968198
- [Derived] Upadhyay P, Joshi A, Mishra I, Kelly L, Novack L, Hariri S, Kveraga K, Subramaniam B. Short Term Effects of Inner Engineering Completion Online Program on Stress and Well-Being Measures. Front Psychol. 2022 Apr 27;13:814224. doi: 10.3389/fpsyg.2022.814224. eCollection 2022. PMID 35572309
- See also: ISHA Foundation Website — https://www.innerengineering.com/ieo-new/completion/